CLINICAL TRIAL: NCT04727723
Title: Two Steps Italian Prospective obsErvationAL Study Assessing the Effectiveness and Outcomes Associated With LUtathera (177Lu) Oxodotreotide Treatment in Adult Subjects With Unresectable or Metastatic, Progressive, Well Differentiated (G1 and G2), Somatostatin Receptor Positive Gastroenteropancreatic-neuroendocrine Tumours (GEP-NETs) - REAL-LU
Brief Title: Italian Prospective Observational Study Assessing the Effectiveness and Outcomes Associated With Lutathera Treatment in GEP-NETs
Acronym: REAL-LU
Status: Active, not recruiting | Type: Observational
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Other Study IDs: CAAA601A0IT02
Record Dates: First submitted 2020-11-20; First posted 2021-01-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
Keywords: GEP-NET; Gastro-Entero-Pancreatic; Neuroendocrine Tumour; AAA; Advanced Accelerator Applications; Luthatera
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lutathera®: Lutathera® will be administered according to the local label and according to the recommended treatment regimen in adults consisting of four equally divided doses of Lutathera® for a total of 29.6 GBq (800 mCi).
  Interventions: Drug: Lutathera®

INTERVENTIONS:
Drug: Lutathera® — Treatment with Lutathera® will be independent from participation in this observational study and must not be initiated for the purpose of participating in this study. The decision to treat patients with Lutathera® will occur before patients are enrolled in the study.

SUMMARY:
This is a multicentre long-term non-interventional study of adult subjects diagnosed with unresectable or metastatic, progressive, well differentiated (G1 and G2), somatostatin receptor positive GEP-NETs who have been prescribed Lutathera® in standard clinical practice.

DETAILED DESCRIPTION:
Data on patients will be collected from the date when patient consent was obtained, during treatment with Lutathera® and for a follow-up period until end of study (EOS), defined as the time when the last enrolled patient has completed 36 months of assessments (unless early termination) after enrolment. Data will be collected in accordance with routine clinical visits.

The study duration will be 48 months in total: 12 months recruitment and 36 of follow-up from the last patient in.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any data collection.
* Patients must be diagnosed with unresectable or metastatic, progressive, well differentiated (G1 and G2), somatostatin receptor positive gastroenteropancreatic-neuroendocrine tumour (GEP-NET).
* Aged ≥18 years.
* Patients must be naïve to treatment with Lutathera® at enrolment.

Exclusion Criteria:

* Participation in a current or prior investigational study within 30 days preceding enrolment or within 5 half-lives of the investigational product, whichever is longer.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll patients with unresectable or metastatic, progressive, well differentiated (G1 and G2), somatostatin receptor positive GEP-NETs.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 48 months
  PFS, defined as the time, in months, from Lutathera® treatment initiation to the date of first objective tumour progression, determined according to Response Evaluation Criteria in Solid Tumours (RECIST) Criteria, Version 1.1, or death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 48 months
  ORR, defined as the proportion of treated patients who achieve a best overall response of partial response (PR) or complete response (CR) according to RECIST 1.1
Duration of Response (DoR), for those patients who achieve a best response of PR or better | Up to 48 months
  DoR, defined as the time, in months, from the date when criteria for response are first met until the date of a progression event (according to the primary definition of PFS).
Clinical Benefit Rate (CBR) | Up to 48 months
  CBR, defined as the proportion of treated patients who achieve a best overall response of stable disease (SD), PR or CR according to RECIST 1.1.
Duration of Clinical Benefit, for those patients who achieve a best response of SD or better | Up to 48 months
  Duration of clinical benefit, defined as the time, in months, from the date when criteria for clinical benefit are first met until the date of a progression event (according to the primary definition of PFS).
Time to Progression (TTP) | Up to 48 months
  TTP, defined as the time, in months, from Lutathera® treatment initiation to the date of first objective tumour progression, assessed according to RECIST 1.1.
Assess the impact of treatment on health-related Quality of Life (HRQoL) by EORTC QLQ-C30 questionnaire | Up to 48 months
  EORTC QLQ-C30 will be filled in by the patient prior to knowing computed tomography (CT) scan/magnetic resonance imaging (MRI) result.
  The EORTC QLQ-C30 questionnaire is designed for use with a wide range of cancer patient populations and is intended to be supplemented by tumour-specific questionnaire modules. The EORTC QLQ-C30 incorporates different multi-item scales, i.e. functional scales, symptom scales and a Global Health Status/QoL scale. All parameters are evaluated using single or multi-item questions which are consequently converted into a 100-point score.
Assess the impact of treatment on health-related Quality of Life (HRQoL) by EORTC QLQ-G.I.NET-21 questionnaire | Up to 48 months
  EORTC QLQG. I.NET-21 will be filled in by the patient prior to knowing computed tomography (CT) scan/magnetic resonance imaging (MRI) result.
  EORTC QLQ-G.I.NET-21 questionnaire is a module specific for neuroendocrine tumours and comprises 21 questions assessing disease symptoms, side effects of treatment, body image, disease related worries, social functioning, communication and sexuality. Each subscale is based on the following items: endocrine scale (items 31-33); gastrointestinal scale (34-38); treatment scale (39, 40, and 46); social function scale (42, 44, and 49); disease related worries scale (41, 43, and 47); muscle/bone pain (48), sexual function (51), information/communication function (50), and body image (45).
  All parameters are evaluated using single or multi-item questions which are consequently converted into a 100-point score
Time to Deterioration (TTD) in global health scale (TTD- global health scale) | Baseline, up to 48 months
  TTD, defined as the time, in months, from Lutathera® treatment initiation to the date of first deterioration of ≥10 points in the EORTC QLQ-C30 and EORTC QLQ-G.I.NET21 global health scale score compared to the baseline score for the same domain.
Time to Deterioration (TTD) in diarrhoea item (TTD- diarrhoea item) | Baseline, up to 48 months
  TTD, defined as the time, in months, from Lutathera® treatment initiation to the date of first deterioration of ≥10 points in the EORTC QLQ-C30 and EORTC QLQ-G.I.NET21 diarrhoea item score compared to the baseline score for the same domain.
Time to Deterioration (TTD) in fatigue item (TTD- fatigue item) | Baseline, up to 48 months
  TTD, defined as the time, in months, from Lutathera® treatment initiation to the date of first deterioration of ≥10 points in the EORTC QLQ-C30 and EORTC QLQ-G.I.NET21 fatigue item score compared to the baseline score for the same domain.
Time to Deterioration (TTD) in pain item (TTD- pain item) | Baseline, up to 48 months
  TTD, defined as the time, in months, from Lutathera® treatment initiation to the date of first deterioration of ≥10 points in the EORTC QLQ-C30 and EORTC QLQ-G.I.NET21 pain item score compared to the baseline score for the same domain.
Number of patients with Adverse Events (AEs) related to study drug | Up to 48 months
  Number of patients with Adverse Events (AEs) related to study drug will be reported
Seriousness and relationship to Lutathera® treatment | Up to 48 months
  Seriousness and relationship to Lutathera® treatment will be reported
Incidence of deaths due to any cause. | Up to 48 months
  Incidence of deaths due to any cause will be reported
Number of participants with notable changes in laboratory parameters | Up to 48 months
  Safety measured by the notable post-baseline changes in laboratory parameters compared to baseline.
  Standard Lab parameters will be reported when performed as clinical practice.
Number of participants with notable changes in physical examination | Up to 48 months
  Safety measured by the notable post-baseline changes in physical examination compared to baseline.
  Physical examination will be reported when performed as clinical practice.
Number of participants with notable changes in vital signs | Up to 48 months
  Safety measured by the notable post-baseline changes in vital signs compared to baseline.
  Vital signs will be reported when performed as clinical practice.
Number of participants with notable changes in electrocardiogram (ECG) | Up to 48 months
  Safety measured by the notable post-baseline changes in ECG compared to baseline.
  ECG results will be reported when performed as clinical practice.
Changes in Karnofsky Performance Status (KPS) scores | Up to 48 months
  KPS scores will be reported when performed as clinical practice. Karnofsky Performance Status (KPS) is a standard way of measuring the ability of cancer patients to perform ordinary tasks. The KPS score ranges from 0 to 100. A higher score means the patient is better able to carry out daily activities. KPS forms must be completed by the treating physician at each treatment and follow-up visit.
Baseline characteristics of patients selected | Baseline
  Baseline characteristics of patients prescribed with Lutathera® (medical and disease history, prior treatments for NETs, baseline and demographic characteristics).
Correlation of possible prognostic factors with clinical effectiveness outcomes. | Up to 48 months
  Potential prognostic factors (e.g., somatostatin receptor (SSTR) expression levels (tumour uptake score) determined by Octreoscan® scintigraphy or 68Ga PET/CT according to clinical practice, standardized uptake value (SUV) of [18F]fluorodeoxyglucose (FDG) PET/CT (if performed), levels of the biomarkers collected in clinical routine, stage of disease at the time of first diagnosis, KPS score at baseline).
Describe radiation emission levels at one metre distance of patients treated | Up to 18 months
  Radiation emission levels at one metre distance of patients treated with Lutathera® at the time of hospital discharge and as collected according to the local Summary of Product Characteristics (SmPC), the "Scheda di Monitoraggio AIFA" and as per clinical practice
Describe dosimetry data after administration (if dosimetry is performed) | Up to 18 months
  Number of patients undergoing dosimetry, dosimetry method used and radiation-absorbed doses to tumour and normal organs after Lutathera® administration.
Number of days of hospitalization for Lutathera® treatment. | Up to 18 months
  Number of days of hospitalization for Lutathera® treatment will be provided
Frequency of hospitalization. | Up to 48 months
  Frequency of hospitalizations will be provided
Duration of hospitalization | Up to 48 months
  Duration of hospitalizations will be provided
Extent of usage of concomitant medications for AE treatment. | Up to 48 months
  Extent of usage of concomitant medications for AE treatment will be provided
Changes in use of concomitant medications for symptoms management | Up to 48 months
  Changes in use of concomitant medications for symptoms management will be provided
Information about the patient's diagnosis-related group (DRG) | Up to 18 months
  Information about the patient's diagnosis-related group (DRG) will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Italy (18):
  - Novartis Investigative Site, Alessandria
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Brescia
  - Novartis Investigative Site, Cona
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Latina
  - Novartis Investigative Site, Meldola
  - Novartis Investigative Site, Messina
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Negrar
  - Novartis Investigative Site, Padua
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Reggio Emilia
  - Novartis Investigative Site, Rionero in Volture
  - Novartis Investigative Site, Roma
  - Novartis Investigative Site, Rozzano
  - Novartis Investigative Site, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lastoria S, Rodari M, Sansovini M, Baldari S, D'Agostini A, Cervino AR, Filice A, Salgarello M, Perotti G, Nieri A, Campana D, Pellerito RE, Pomposelli E, Gaudieri V, Storto G, Grana CM, Signore A, Boni G, Dondi F, Simontacchi G, Seregni E. Lutetium [177Lu]-DOTA-TATE in gastroenteropancreatic-neuroendocrine tumours: rationale, design and baseline characteristics of the Italian prospective observational (REAL-LU) study. Eur J Nucl Med Mol Imaging. 2024 Sep;51(11):3417-3427. doi: 10.1007/s00259-024-06725-7. Epub 2024 May 22. PMID 38772998